CLINICAL TRIAL: NCT06286865
Title: Improving Quality of ICD-10 (International Statistical Classification of Diseases, Tenth Revision) Coding Using AI: Protocol for a Crossover Randomized Controlled Trial
Brief Title: Improving Quality of ICD-10 Coding Using AI: Protocol for a Crossover Randomized Controlled Trial
Acronym: ClinCode
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Taridzo Chomutare, Senior Researcher, University Hospital of North Norway
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 260972(REK)
Record Dates: First submitted 2024-02-16; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Gastrointestinal Diseases
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Easy-ICD interface (Active Comparator): This arm uses our AI-based computer-assisted clinical coding (CAC) system, Easy-ICD
  Interventions: Other: Easy-ICD
- Control interface (No Intervention): This control arm uses an interface similar to Easy-ICD, but without the AI functionality

INTERVENTIONS:
Other: Easy-ICD — Easy-ICD is an AI-based computer-assisted clinical coding (CAC) system that helps clinical coder assign ICD-10 codes to clinical notes such as discharge summaries.
  Arms: Easy-ICD interface

SUMMARY:
The goal of this randomised trial is to learn about the role of AI in clinical coding practice. The main question it aims to answer is:

Can the AI-based CAC system reduce the burden of clinical coding and also improve the quality of such coding? Participants will be asked to code clinical texts both while they use our CAC system and while they do not.

DETAILED DESCRIPTION:
Once participants are recruited, they are randomly allocated to 2 groups without allocation concealment. Allocation concealment will not be relevant for clinical coders since it is known whether a participant is assisted or not, and we will not develop a placebo coding assistant. We will, however, conceal the allocation of subjects for the analyses.

In total, participants will code 20 clinical notes, where each note belongs to a single patient. The participants are asked to complete the experiment in 1 sitting without interruptions, and they cannot revisit or go back to previous notes. In the event that participants are interrupted, they are asked to exit the experiment, and any incomplete records are discarded as invalid.

The user study process can be summarized in the following steps:

1. Study participants are randomly allocated to group 1 and group 2.
2. To prepare participants for the experiment, a short video tutorial is played after the consent form is signed and right before the clinical coding task commences.
3. In period 1 with 10 clinical notes, group 1 uses the control interface, while group 2 uses the intervention interface.
4. Data are logged in the background using button presses (eg. time, assigned codes, and comments).
5. Then, there is an immediate crossover to period 2 for the last 10 clinical notes.
6. Data continue to be logged in the background using button presses.
7. At the end, participants in both groups will complete the system usability scale.

ELIGIBILITY:
Inclusion Criteria:

* participant has coded clinical texts before, preferably ICD-10 coding
* is a healthcare professional, eg. clinician, nurse, professional coders
* can understand Swedish

Exclusion Criteria:

* participants outside Norway and Sweden

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Time | 1 hour
  Time in seconds taken to assign ICD-10 codes to each of the 20 clinical notes.
Accuracy | 1 hour
  Accuracy is calculated by dividing the number of correct ICD-10 codes by the total number of codes assigned.

CONTACTS AND LOCATIONS:
Overall Officials: Hercules Dalianis, PhD, Principal Investigator — Norwegian Centre for E-health Research
Locations (1):
- Norwegian Centre for E-health Research, Tromsø, Troms, Norway

IPD SHARING:
Plan to Share IPD: Yes
The data we collect in the study are all anonymous and will be shared publicly after the user study is published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the publishing of the user study.
Access Criteria: The anonymous data will be publicly available.

REFERENCES:
- [Derived] Chomutare T, Lamproudis A, Budrionis A, Svenning TO, Hind LI, Ngo PD, Mikalsen KO, Dalianis H. Improving Quality of ICD-10 (International Statistical Classification of Diseases, Tenth Revision) Coding Using AI: Protocol for a Crossover Randomized Controlled Trial. JMIR Res Protoc. 2024 Mar 12;13:e54593. doi: 10.2196/54593. PMID 38470476